CLINICAL TRIAL: NCT03536767
Title: An Open-Label Extension and Safety Monitoring Study of Patients with Symptomatic Transthyretin Cardiomyopathy Who Have Completed the Phase II Study AG10-201
Brief Title: Open-Label Study of AG10 in Patients with Cardiomyopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG10-202
Record Dates: First submitted 2018-05-11; First posted 2018-05-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Amyloid Cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label (Experimental)
  Interventions: Drug: AG10

INTERVENTIONS:
Drug: AG10 — AG10 800mg twice daily, oral administration
  Other Names: TTR Stabilizer

SUMMARY:
This prospective, multicenter open-label study will evaluate the long-term safety, tolerability, PK and PD of AG10 administered on a background of stable heart failure therapy.

DETAILED DESCRIPTION:
An Open-Label Extension and Safety Monitoring Study of Patients with Symptomatic Transthyretin Cardiomyopathy Who Have Completed the Phase II Study AG10-201

The primary objective of this study is to evaluate the long-term safety and tolerability of AG10 administered to adult patients with symptomatic transthyretin amyloid cardiomyopathy (ATTR-CM) in patients who have completed the study AG10-201.

This study will be an Open-Label Extension and Safety Monitoring Study of up to 55 male and/or female patients with symptomatic ATTR-CM aged 18 through 90 years, who have completed the Phase II Study AG10-201. Enrollment into the study will be followed by visits at Day 14, Day 45, 3 Months and every 3 months thereafter until Month 54. After the Month 54 Visit, study visits will be every 6 months. There will be one follow-up visit approximately 30 days after last dose.

If all doses are well tolerated, the duration of each patient's participation in the study will continue based on periodic recommendations of the AG10 Data Monitoring Committee (DMC) and/or registration of the product for the treatment of symptomatic ATTR-CM.

The secondary objectives of this study are to characterize the pharmacokinetics (PK) of AG10 administered orally twice daily in patients with symptomatic ATTR-CM, and to describe the long-term pharmacodynamic (PD) properties of AG10 as assessed by established assays of transthyretin (TTR) stabilization, including Fluorescent Probe Exclusion (FPE) assay and Western blot, and to describe the PK-PD relationship of AG10 in adult patients with symptomatic ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

1. Completed participation in study AG10-201.
2. Willing and able to comply with the study medication regimen and all study requirements.
3. The ability to understand and provide informed consent, which must be obtained prior to initiation of study participation.
4. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use effective method(s) of contraception.

Exclusion Criteria:

1. Hemodynamic instability that would pose too great a risk to the subject.
2. Abnormalities in clinical laboratory tests that would pose too great a risk to the subject.
3. Any clinically significant ongoing medical condition or any laboratory abnormality or condition that could adversely affect the safety of the patient.
4. Known hypersensitivity to study drug (AG10), its metabolites, or formulation excipients.
5. Likely to undergo heart transplantation or placement of a mechanical circulatory device within the next year.
6. Receiving current treatment with diflunisal, tafamidis, green tea, doxycycline, TUDCA/Ursodiol, patisiran, inotersen or any other investigational ATTR agent within 14 days or 5 half-lives of the prior investigational agent (whichever is longer) prior to dosing with study drug.
7. Females who are pregnant or breastfeeding. Lactating females must agree to discontinue nursing before the study drug is administered.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of long-term safety and tolerability: Incidence of each treatment-emergent adverse events | up to 60 Months or study completion by recommendation from safety monitoring committee
  Incidence of each treatment-emergent adverse events

SECONDARY OUTCOMES:
AG10 Pharmacokinetics AUC | up to 60 Months or study completion by recommendation from safety monitoring committee
  Area under the plasma concentration-time curve (AUC)
AG10 Pharmacodynamic Assessments of TTR stabilization by Fluorescent Polarization Exclusion Assay | up to 60 Months or study completion by recommendation from safety monitoring committee
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays: Fluorescent Polarization Exclusion Assay (FPE)
AG10 Pharmacodynamic Assessments of TTR stabilization by Western Blot | up to 60 Months or study completion by recommendation from safety monitoring committee
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays: Immunoblotting (Western Blot)
AG10 Pharmacodynamic Assessments: prealbumin | up to 60 Months or study completion by recommendation from safety monitoring committee
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays: quantitation of prealbumin (TTR).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No